CLINICAL TRIAL: NCT00341614
Title: The Effects of an Exercise and Diet Intervention on Cardiovascular Risk Factors in Postmenopausal Type 2 Diabetics
Brief Title: Exercise Training in Older Diabetic Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of San Francisco (Other)
Collaborators: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FDF-05-06
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2007-08-16 (Estimated); Status verified 2007-08

CONDITIONS: Cardiovascular Diseases; Diabetes Mellitus, Type 2
Keywords: Exercise; Diabetes Mellitus, Type 2; Postmenopause; Diet
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus, Type 2; Motor Activity | interventions — Exercise; Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: 3-month Exercise Training and Diet Education

SUMMARY:
Type 2 diabetics (non-insulin-dependent) are more than five times as likely to suffer an initial myocardial infarction (MI; heart attack) compared to nondiabetics.Female diabetics in particular, have a higher mortality rate for coronary artery disease (CAD) than male diabetics.C-reactive protein measurement in the clinical setting enhances the detection of individuals who are at high risk for cardiovascular disease (CVD), by providing additional predictive value.

We propose to study the effects of a supervised exercise and diet intervention on cardiovascular disease risk in postmenopausal diabetic women. We will recruit 35 postmenopausal, sedentary type 2 diabetics who will undergo a 3 month exercise and dietary intervention. They will exercise 3 times a week for 30 min in a supervised setting. Exercise mode will be aerobic and self-selected (i.e. treadmill, bike) at an intensity level of 50-85% VO2peak. Blood glucose will be monitored before and after exercise. The dietary intervention will consist of 6 meetings with a registered dietitian.

The study is designed to test the following hypotheses:

* Cardiovascular disease risk measures will be different following a 3-month exercise and diet intervention.

  * H1: Blood markers for coronary artery disease risk, as measured by CRP, TC, LDL, TG, FG, fasting insulin, and HbA1c, will be different following a 3-month exercise and diet intervention.
  * H2: Anthropometric measures of coronary artery disease risk, as measured by WHR, will be different following a 3-month exercise and diet intervention.
  * H3: Resting blood pressure, as measured by SBP and DBP, will be different following a 3-month exercise and diet intervention.
  * H4: Total body fat, as measured by DXA, will be different following a 3-month exercise and diet intervention.
* Health-related measures will be different following a 3-month exercise and diet intervention.

  * H1: Cardiorespiratory fitness, as measured by maximal oxygen consumption (VO2max) will be different following a 3-month exercise and diet intervention.
  * H2: Bone-mineral density, as measured by DXA, will be different following a 3-month exercise and diet intervention.
  * H3: Dietary measures (total daily kcal, and daily fat kcal) will be different following a 3-month exercise and diet intervention.

DETAILED DESCRIPTION:
* Recruitment: Participants who have signed up for the research recruitment mailing list at the UCSF/Mt. Zion Osteoporosis Center will be mailed a CHR approved recruitment letter that briefly describes the study purpose and eligibility criteria. Only the individual's name and address are on the mailing list; there is no medical information. Medical records are not accessed. Telephone screening will take place in the ESS Department at USF. A script will be followed.
* Pre and Post-Testing: Interested subject candidates will be scheduled to meet with Dr. Orri or Dr. Thompson at USF to provide written informed consent and complete a health history questionnaire (see appendix) to evaluate their CV risk. They will obtain written medical notification from their physician stating that they are in adequate diabetic control and cleared to begin an exercise program. Once selected, measurements of HT, WT, WHR, SBP, and DBP will take place in the ESS lab at USF.
* Blood draws: Subjects will arrive at the UCSF GCRC after a 12-hr fast. The blood variables obtained will include: CRP, TC, LDL-C, HDL-C, TG, FG, fasting insulin (HOMA calculated for marker of insulin resistance), and HbA1c. Approximately 2 tablespoons of blood will be drawn.
* Bone mineral density: BMD measurements (dual X-ray absorptiometry, DXA) will take place at the General Clinical Research Center at UCSF following the blood draw. A snack will be provided to the subjects prior to entering the DXA scanning area.
* Cardiorespiratory fitness: Maximal exercise testing will be using a treadmill protocol in the Exercise Physiology Laboratory at UCSF General Clinical Research Center. Tests will be conducted by Dr. Orri, Dr. Thompson, and Joanne Krasnoff, M.S. The Naughton protocol will be used in which the grade is increased 3.5% every 2 min, while the speed remains at 2 mph after the warmup. The subject continues until volitional exhaustion or the exercise technicians terminate test end as designated by the American College of Sports Medicine (ACSM).

All participants will have a 12-lead electrocardiogram (ECG) during the testing sessions to monitor for dysrhythmias or ischemia. Heart rate and blood pressure will be monitored every 2 minutes. Rating of perceived exertion (RPE) will be assessed every minute of the test. Maximal oxygen uptake (VO2max), as well as maximal levels of blood pressure, heart rate, respiratory exchange ratio (RER), and RPE will be recorded at the end of the test and used to determine the exercise training intensity. Expired gases will be collected throughout the test with CO2 and O2 and volume analyzed for calculation of oxygen uptake using a Quinton QMC computerized gas analysis system (Quinton Instruments, Bothell WA). All exercise technicians will be CPR and first-aid certified.

* Body composition and BMD: Per cent body fat (%BF) and BMD will determined using dual energy X-ray absorptiometry (DXA). All scans will be done on a GE-Lunar Prodigy (Madison, WI). Variables of interest from the DXA scan will be %BF, total fat mass, lean body mass (LBM), and bone mineral density in g/cm2.
* Exercise intervention: The 3-month exercise intervention will take place at the Millberry Union fitness center at UCSF, times per week for 30 min each session, accompanied by certified fitness professional who is trained to work with special populations. All standard emergency procedures will be followed by the trained UCSF staff.
* Exercise program design: Study participants will be required to complete 36 exercise sessions in the 12 week program. They will exercise a minimum of 3 times per week for 30 min, accompanied by certified fitness professional who is trained to work with special populations. Participants will wear a HR monitor and be instructed to maintain an intensity in the range of 50-85% VO2peak obtained through max testing. During the initial phase of training (first 4 weeks), participants who are unable to exercise continuously for 30 minutes will perform intermittent exercise bouts of 10 minutes followed by 5 min of rest. Mode of exercise will be self-selected and will involve large muscle groups, incorporating any combination of the following machines: treadmill, stationary cycle, elliptical, Stairmaster, or rowing ergometer.
* Blood glucose monitoring: Participants will be instructed to consume a snack 30-60 min before exercise. Prior to beginning each exercise session, all subjects will monitor their blood glucose to verify that it is between 100 and 250 mg/dl, in the absence of hypo/hyperglycemic symptoms (6). In addition, subjects will be monitored for 30 min post-exercise to verify that their BG is > 70 mg/dl. Juice and protein snacks (peanut butter & crackers) will be available to the subjects in case of post-exercise hypoglycemia. The exercise supervisor will be aware of those subjects who are taking medications that promote insulin production and will carry a glucagon pen. Late-evening exercise sessions will be avoided in order to prevent nocturnal hypoglycemia.
* Dietary intervention: The subjects will receive six 30-min nutrition group counseling sessions with a dietitian. Sessions 1 and 6 will involve instruction on preparing 3-day dietary logs, while sessions 2-5 will consist of selected topics (i.e. dietary recommendations, low sodium diets, blood glucose control).

ELIGIBILITY:
Inclusion Criteria:

* Female 45-75 yrs old
* Type 2 diabetic for > 6 months
* "Reasonable" control of diabetes

  * blood glucose within 100-250 mg/dl prior to exercise
  * absence of hypoglycemic symptoms
  * diabetes control verified by physician
  * cleared by physician to begin exercise program
* Postmenopausal > 6 months
* Sedentary
* Ability and willingness of patient to give written, informed consent
* Able and willing to participate in an exercise intervention

Exclusion Criteria:

* Diabetes not in control

  * unable to maintain blood glucose within 100-250 mg/dl
  * development of urinary ketone bodies (ketosis)
  * symptoms of hypoglycemia before, during, and post-exercise
  * no physician's approval to participate
* Male
* Female <45 or >75 yr
* > 300 lb (weight limit for DXA table)
* On insulin
* Contraindications to Exercise Testing (ACSM, 2000)
* Ischemia
* Recent myocardial infarction
* Unstable angina
* Uncontrolled cardiac arrhythmias
* Severe aortic stenosis
* Uncontrolled heart failure
* Acute pulmonary embolus
* Acute myocarditis or pericarditis
* Dissecting aneurysm
* Acute infections
* Electrolyte abnormalities
* Severe hypertension (SBP > 200 mm Hg, DBP > 110 mm Hg at rest)
* Tachyarrhythmias or bradyarrhythmias
* Hypertrophic cardiomyopathy
* Neuromuscular, musculoskeletal, or rheumatoid disorders that are exacerbated by exercise
* Not able to complete exercise testing (i.e must be ambulatory and without orthopedic limitations which would preclude maximal effort exercise)

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2006-06; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
VO2max at 3 months | 3 months
C-reactive protein at 3 months | 3 months
Blood lipids (total cholesterol, LDL, HDL, TC/HDL ratio, triglycerides) at 3 months | 3 months
Fasting glucose at 3 months | 3 months
Fasting insulin (insulin resistance) at 3 months | 3 months
HbA1C at 3 months | 3 months
Body fat % at 3 months | 3 months
Blood pressure (SBP, DBP) at 3 months | 3 months
Waist-hip ratio at 3 months | 3 months
Total kcal and fat kcal at 3 months | 3 months

SECONDARY OUTCOMES:
Bone-mineral density at 3 months | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Sellmeyer, M.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States